CLINICAL TRIAL: NCT05184049
Title: Effects of Epalrestat on Peripheral Neuropathy and Central Nervous System in Diabetic Patient
Brief Title: Effects of Epalrestat on Peripheral Neuropathy and Central Nervous System in Diabetic Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiangya Hospital of Central South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20210406
Record Dates: First submitted 2021-11-02; First posted 2022-01-11 (Actual); Last update posted 2022-01-11 (Actual); Status verified 2021-10

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — epalrestat; mecobalamin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Epalrestat (Experimental): oral epalrestat (50mg/ time, 3 times/day) + conventional hypoglycemia + oral mecobalamin (0.5mg/ time, 3 times/day) for half a year
  Interventions: Drug: Epalrestat,Mecobalamin
- The control group (Experimental): conventional hypoglycemia + oral mecobalamin (0.5mg/ time, 3 times/day) for half a year
  Interventions: Drug: Mecobalamin

INTERVENTIONS:
Drug: Epalrestat,Mecobalamin — Epalrestat will be taken orally at a dose of 50mg 3 times a day before meals. In addition, conventional hypoglycemic and oral mecobalamin treatment 0.5mg/ time, 3 times/day, before meals.
  Arms: Epalrestat
Drug: Mecobalamin — Subjects takes mecobalamin 0.5mg orally, 3 times a day.Regular hypoglycemia.
  Arms: The control group

SUMMARY:
This study evaluated the efficacy of epalrestat in diabetic peripheral neuropathy and its effects on the central nervous system in diabetic peripheral neuropathy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged 18 to 65 years (to the date of screening)；
2. A clear history of type 2 diabetes (using the 1999 WHO diabetes diagnostic criteria) with a course of disease > 6 months;
3. HbA1c < 7%;
4. Two or more of the following five tests are abnormal: abnormal temperature perception; Nylon wire for hypoesthesia or disappearance of the foot; Abnormal vibration sense; Ankle reflex disappeared; Two or more nerve conduction velocities were reduced;
5. Have not used mecobalamin, epalrestat, lipoic acid or high-dose glucocorticoid in the recent (3 months) period, or have not been involved in other treatment of the same disease within 3 months prior to the study;

Exclusion Criteria:

1. Neuropathy caused by other causes, such as cervical and lumbar lesions, cerebral infarction, etc.;
2. With acute metabolic complications of diabetes, such as ketoacidosis, lactic acidosis, diabetes hyperotonic state, etc;
3. Severe cardiovascular and cerebrovascular diseases , pulmonary heart disease or pulmonary insufficiency, renal failure, severe dyslipidemia, poorly controlled hypertension, severe hepatitis.
4. Those with a history of malignant tumor or wasting diseases such as tuberculosis;
5. Contraindications to MRI scanning: such as internal (especially oral) metal implants, claustrophobia, etc;
6. Poor compliance or serious side effects;
7. pregnant female.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2022-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
The change of resting-state functional Magnetic Resonance Imaging | baseline , 6months
  The change in grey matter volume,white matter area, local gyrification index after 6-months treatment

SECONDARY OUTCOMES:
Mean change of electromyography | baseline , 6months
  mean change from baseline in nerve conduction velocity(m/s) after 6-months treatment
Mean change of quantitative somatosensory testing | baseline , 6months
  Mean change of temperature perception threshold(℃) after 6-months treatment
Mean change of corneal confocal focus | baseline , 6months
  Mean change of nerve fibre density(no./mm2) after 6-months treatment
Mean change in HbA1c | baseline , 6months
  Mean change of HbA1c(%) after 6-months treatment
Change of Self-Rating Anxiety Scale | baseline , 6months
  Mean change of Self-Rating Anxiety Scale score after 6-months treatment score.The minimum and maximum values is 25 and 100, which higher scores mean more anxiety.
Change of Self-Rating Depression Scale | baseline , 6months
  Mean change of Self-Rating Depression Scale score after 6-months treatment.The minimum and maximum values is 25 and 100, which higher scores mean more depression.
Mean change of Toronto clinical scoring system | baseline , 6months
  Mean change of Toronto clinical scoring system score after 6-months treatment.The minimum and maximum values is 0 and 19, which higher scores mean more severe neuropathy.
Mean change of Neuropathic pain scale | baseline , 6months
  Mean change of Neuropathic pain scale score after 6-months treatment.The minimum and maximum values is 0 and 10, which higher scores mean more severe neuropathy.
Mean change of Michigan neuropathy screening form | baseline , 6months
  Mean change of Michigan neuropathy screening form score after 6-months treatment.The minimum and maximum values is 0 and 23, which higher scores mean more severe neuropathy.
Mean change of mini-mental state examination | baseline , 6months
  Mean change of mini-mental state examination score after 6-months treatment.The minimum and maximum values is 0 and 30, which lower scores mean more severe cognitive dysfunction.
Mean change of Montreal Cognitive Assessment | baseline , 6months
  Mean change of Montreal Cognitive Assessment score after 6-months treatment.The minimum and maximum values is 0 and 30, which lower scores mean more severe cognitive dysfunction.

CONTACTS AND LOCATIONS:
Locations (1):
- Xiangya Hospital of Central South University, Changsha, Hunan, China